CLINICAL TRIAL: NCT04520295
Title: Predictive Biomarkers Screening by ctDNA Detection in Advanced HER2 Positive Gastric Cancer Patients Treated by Trastuzumab Plus Chemotherapy
Brief Title: ctDNA Screening in Advanced HER2 Positive Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhang, Chair of Department of Oncology, Ruijin Hospital
Other Study IDs: BSctDNA-GC
Record Dates: First submitted 2020-08-06; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: HER2-positive Gastric Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HER2 positive cohort
  Interventions: Genetic: ctDNA screening

INTERVENTIONS:
Genetic: ctDNA screening — Molecular events including gene mutation, fusion and amplification will be detected by next generation sequencing platform (OncoScreen Plus panelTM) using ctDNA collected from peripheral blood samples of gastric cancer patients. For HER2 positive patients, samples will be collected at baseline, first surveillance after treatment and disease progression. For HER2 negative patients, samples will be collected at baseline as negative control.

SUMMARY:
To identify molecular biomarker panel correlating with efficacy of trastuzuamb in advanced HER2 positive gastric cancer patients. To observe the molecular evolution of HER2 positive gastric cancer during treatment by ctDNA detection.

DETAILED DESCRIPTION:
Molecular events including gene mutation, fusion and amplification will be detected by next generation sequencing platform (OncoScreen Plus panelTM) using ctDNA collected from peripheral blood samples of gastric cancer patients. For HER2 positive patients, samples will be collected at baseline, first surveillance after treatment and disease progression. For HER2 negative patients, samples will be collected at baseline as negative control.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patients aged over 18 years.
2. Histologically confirmed gastric adenocarcinoma. Gastric tumors should be treatment naïve unresectable or metastatic disease, or recurrence over 6 months after finish of adjuvant chemotherapy.
3. HER2 status is confirmed by IHC/FISH. HER2 positive: IHC 3+ or IHC 2+ plus FISH positive, HER2 negative: IHC 0/1+ or IHC 2+ plus FISH negative.
4. At least one measurable lesion should be confirmed by imaging examination.
5. Eligible peripheral blood samples
6. Patients with enough organ function and performance status (ECOG 0-2) can tolerant chemotherapy.
7. For HER2 positive patients, trastuzumab should be used as first-line treatment. The regimen of chemotherapy should be platinum plus oral fluorouracil.
8. For HER2 negative patients, clinicopathological characteristics should be matched to HER2 positive patients.
9. Willing to provide clinicopathological information and imaging information.

Exclusion Criteria:

1. Patients received systemic treatment before enrolled or finished adjuvant chemotherapy less than 6 months.
2. With second primary malignant diseases.
3. Other situations assessed by investigator can disturb quality control of the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2 positive gastric cancer patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-19 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in molecular biomarkers at time on best overall response | 36 months
  Molecular biomarkers including gene mutation, amplification and fusion were detected by next generation sequencing platform (OncoScreen Plus panelTM) using ctDNA collected from patients during treatment. The list of genes included in OncoScreen Plus panelTM is provided as supplementary file.

SECONDARY OUTCOMES:
Change from baseline in molecular biomarkers at time on disease progression | 36 months
  Molecular biomarkers including gene mutation, amplification and fusion were detected by next generation sequencing platform (OncoScreen Plus panelTM) using ctDNA collected from patients during treatment. The list of genes included in OncoScreen Plus panelTM is provided as supplementary file.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Principal Investigator — Ruijin Hospital
Locations (1):
- Department of Oncology, Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No